CLINICAL TRIAL: NCT00640588
Title: Prospective Exploratory Study to Describe in CHB naïve and Non-naïve Patients, Hepatitis B Virus (HBV) Kinetics During the First 24 Weeks of Treatment With Telbivudine
Brief Title: Prospective Exploratory Study to Describe Hepatitis B Virus (HBV) Kinetics During Treatment With Telbivudine
Acronym: EBEREST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLDT600AES01
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, chronic; Viral kinetics; Telbivudine; Adefovir; Compliance
MeSH Terms: conditions — Hepatitis B, Chronic; Patient Compliance | interventions — Telbivudine; adefovir dipivoxil; adefovir

ARMS (2):
- 1 (Experimental): Telbivudine
  Interventions: Drug: Telbivudine
- 2 (Active Comparator): Arm 2: 600 mg/day, oral telbivudina plus 10 mg/day oral adefovir for 24 weeks
  Interventions: Drug: oral adefovir

INTERVENTIONS:
Drug: Telbivudine — Arm 1: 600 mg/day, oral telbivudina for 24 weeks
  Other Names: Sebivo; Tyzeka; Hepsera
  Arms: 1
Drug: oral adefovir — Arm 2: 600 mg/day, oral telbivudina plus 10 mg/day oral adefovir for 24 weeks
  Other Names: adefovir
  Arms: 2

SUMMARY:
This study will explore HBV kinetics in CHB patients during the first 24 weeks of treatment with telbivudine

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Documented compensated HBeAg negative CHB defined by baseline HBV serology, DNA and ALT criteria.

Exclusion Criteria:

* Co-infection with HCV, HDV, or HIV.
* Prior therapy with nucleos(t)ides in NAÏVE patient and prior treatment with lamivudine in patients with suboptimal response to adefovir.
* History of hepatic decompensation
* History of malignancy
* Patient has one or more additional known primary or secondary causes of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HBV viral load will be measured by HBV DNA quantification in plasma (log opies/mL) at baseline, 2, 4, 8, 12, 16, 20 and 24 weeks | at baseline, 2, 4, 8, 12, 16, 20 and 24 weeks

SECONDARY OUTCOMES:
Liver function assessed at baseline, 2, 4, 8, 12, 16, 20 and 24 weeks HBV genotype measured at baseline | at baseline, 2, 4, 8, 12, 16, 20 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Barcelona, Spain